CLINICAL TRIAL: NCT07222306
Title: Investigating the Therapeutic Impact of Cannabinoids on Neuroinflammation and Neurobiological Underpinnings of Suicide Ideation in Veterans With PTSD
Brief Title: Cannabis, Neuroinflammation, and Suicidal Ideation: A Supplemental Brain Imaging Study
Acronym: CNS
Status: Enrolling by invitation | Type: Observational
Sponsor: Wayne State University (Other)
Collaborators: Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Principal Investigator, Hilary Marusak, Associate Professor, Wayne State University
Other Study IDs: IRB-24-09-7226; VMR2022-02 (Other Grant/Funding Number: State of Michigan)
Record Dates: First submitted 2025-10-24; First posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: PTSD; Suicidal Thoughts and Behaviors; PTSD Symptoms; Depressive Symptoms
Keywords: PTSD; Suicidal Thoughts; Cannabis; Brain Imaging; MRI; PET; Veterans; Depression; Cannabidiol; THC
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Suicidal Ideation; Behavior; Depression; Marijuana Abuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PET and/or MRI: Positron emission tomography (PET) imaging with the radiotracer, 1-(2-[+F]fluoroethyl)-L-tryptophan or [18F]FETrp and/or magnetic resonance imaging (MRI)
  Interventions: Drug: 1-(2-[+F]fluoroethyl)-L-tryptophan

INTERVENTIONS:
Drug: 1-(2-[+F]fluoroethyl)-L-tryptophan — 1-(2-[+F]fluoroethyl)-L-tryptophan tracer will be used during PET imaging

SUMMARY:
This study will be the first to use brain imaging to explore how cannabis affects the brain and inflammation in U.S. military veterans with PTSD. It builds on an ongoing study testing different combinations of THC and CBD in 200 veterans. In this project, up to 100 veterans will complete brain scans before and after 12 weeks of cannabis administration to see how the brain changes over time. The scans will measure a marker sensitive to neuroinflammatory state, brain communication, and activity during thinking and emotion tasks. By linking these brain changes to improvements in PTSD symptoms, suicidal thoughts, and quality of life, this study may help identify which veterans benefit most from cannabis-based treatments and support more personalized care for PTSD.

DETAILED DESCRIPTION:
This study, referred to here as the 'Neuroimaging Study,' is a supplement (add-on) to our ongoing VMR study (Wayne State Warriors Marijuana Clinical Research Program: Investigating the Impact of Cannabinoids on Veterans' Behavioral Health", PIs: Lundahl and Ledgerwood), which will be referred to as the 'Parent Study'. The Neuroimaging Study will be the first-ever neuroimaging study of cannabis treatment in US armed forces veterans with PTSD, or in any population. The Parent Study involves randomizing 200 veterans with PTSD into one of four different THC (∆9-tetrahydrocannabinol) : CBD (cannabidiol) dose conditions (High THC:High CBD; HighTHC:Low CBD; Low THC:High CBD, and Low THC:Low CBD) for a 12-week treatment phase. For the Neuroimaging Study, half of the 200 participants from the Parent Study (up to N=100; i.e., roughly 25 of the 50 participants in each dose condition) will additionally complete two brain imaging assessments: one before (i.e., 'baseline' scan) and one after the 12-week treatment period (i.e., 'post-treatment' scan). Primary outcomes include: A) neuroinflammatory state as measured via positron emission tomography (PET) imaging with the radiotracer, 1-(2-[+F]fluoroethyl)-L-tryptophan or [18F]FETrp; B) resting or 'basal' neural network communication as measured via functional magnetic resonance imaging (fMRI); and C) brain activation during well-validated inhibitory control (Go/No-Go), emotion regulation (Emotional Stroop), and reward processing (Duke Card Guessing) tasks as measured via fMRI. We will focus on brain regions that are consistently linked to both PTSD symptom severity and suicidal ideation, and that are densely populated with cannabinoid receptors (which are modulated by acute cannabis/cannabinoid administration). Further, the collection of whole-brain, multi-modal neuroimaging data (structural MRI, functional MRI, and PET imaging data) during the same session will allow us to explore the impact of cannabis/cannabinoid administration on the relationship between neuroinflammatory state and neural network activation and interactions throughout the brain, and link these brain metrics to clinical outcomes (e.g., reduction in suicidal ideation or PTSD/depression symptoms over time). This highly innovative approach will provide unprecedented insight into the neurobiological underpinnings of PTSD and suicidal ideation and the potential therapeutic effects of cannabis (and associated brain mechanisms) on these and other critical outcomes (e.g., quality of life, depressive symptoms). Findings from this Neuroimaging Study may also identify veterans who will benefit most from cannabinoid therapeutics and specific THC:CBD dose combinations therein, and thus, may inform a personalized medicine approach for veterans with PTSD in the future.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for, and provided written informed consent to participate in, the Parent Study (NCT06381180) and to be contacted regarding 'future research studies.'
* Able/willing to provide written informed consent to participate in the Neuroimaging Study.

Exclusion Criteria (eligible if the subject does not meet both criteria):

* Contraindications for MRI scanning include, but are not limited to: as braces, pacemaker, implanted metal (self-report MR screening form and ferromagnetic detectors) or medical conditions that prevent comfortable MRI scanning procedures, e.g., inability to lay supine for 60 minutes, claustrophobia, or body weight > 275lbs.
* Contraindications for PET [18F]FETrp imaging include, but are not limited to: chronic medical conditions that alter radiotracer pharmacokinetic properties, e.g, Diabetes I/II (or uncontrolled glucose levels [>200mg/dl non-fasting]), abnormal BMI (<18.5 or > 35kg/m2), autoimmune diseases, or other chronic inflammatory conditions, or take medications (3+ days/week) that will alter radiotracer binding, e.g., glucose stabilizing medications, proton-pump inhibitors, or anti-inflammatory agents, or have medical conditions that prevent comfortable PET scanning procedures, e.g., inability to lay supine for ~75 minutes, tolerate a radial vein catheter and up to 35ml of whole blood drawn, or body weight > 275lbs.

Ages: 19 Years to 69 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — Females must not be pregnant
Study Population: Military veterans with PTSD
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2030-08-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
[18F]FETrp K-complex | Baseline and follow-up (at least 12 weeks after baseline)
  To quantify kynurenine uptake rate, a Patlak graphical analysis will be performed using the image-derived input function and the dynamic brain emission data. This method yields the unidirectional uptake rate constant, K-complex, in each brain region of interest. Outcome analyses will investigate associations with clinical symptoms and cognitive function at baseline, as longitudinal changes from baseline to follow-up with inter-group differences between dose conditions of particular interest.
BOLD fMRI response | Baseline and follow-up (at least 12 weeks after baseline)
  BOLD fMRI response will be isolated by contrasting activation to the contrast Go/No-Go > Rest for the inhibitory control task, iI > cI for the emotion regulation task, and reward > loss for the reward task.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Woodcock, Principal Investigator — Wayne State University; Hilary Marusak, PhD, Principal Investigator — Wayne State University
Locations (1):
- Tolan Park Medical Building, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Etkin A, Prater KE, Hoeft F, Menon V, Schatzberg AF. Failure of anterior cingulate activation and connectivity with the amygdala during implicit regulation of emotional processing in generalized anxiety disorder. Am J Psychiatry. 2010 May;167(5):545-54. doi: 10.1176/appi.ajp.2009.09070931. Epub 2010 Feb 1. PMID 20123913
- [Background] Fonzo GA, Etkin A, Zhang Y, Wu W, Cooper C, Chin-Fatt C, Jha MK, Trombello J, Deckersbach T, Adams P, McInnis M, McGrath PJ, Weissman MM, Fava M, Trivedi MH. Brain regulation of emotional conflict predicts antidepressant treatment response for depression. Nat Hum Behav. 2019 Dec;3(12):1319-1331. doi: 10.1038/s41562-019-0732-1. Epub 2019 Sep 23. PMID 31548678